Official Title: Improving Care Coordination for Adolescents and Young Adults With Cancer:

Implementing a Bridge Between Needs and Services

NCT04586127

IRB-Approved Date: 12/16/21



Social Sciences and Health Policy

# IMPROVING CARE COORDINATION FOR ADOLESCENTS AND YOUNG ADULTS WITH CANCER: IMPLEMENTING A BRIDGE BETWEEN NEEDS AND SERVICES

Informed Consent Form to Participate in Research <u>Sarah Birken, PhD</u>, Principal Investigator Emily Haines, PhD, Co-investigator

#### **SUMMARY**

You are invited to participate in a research study. The purpose of this research is to seek feedback on an intervention designed to assess and address the needs of adolescents and young adults (AYAs) with cancer: the AYA Needs Assessment & Service Bridge (NA-SB). You are invited to be in this study because you a provider serving AYAs with cancer. Your participation in this research will involve participating in a 60-minute telephone interview.

Participation in this study will asking you questions about how NA-SB might be implemented at your institution. All research studies involve some risks. A risk to this study that you should be aware of is a slight risk of breach in confidentiality, although we will take measures to protect your privacy. You will not directly benefit from your participation in this study, but your feedback on NA-SB will help us to refine it so that it better addresses the needs of AYAs and cancer care providers.

Your participation in this study is voluntary. You do not have to participate in this study if you do not want to. You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. The person in charge of this study is Sarah Birken, PhD. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his/her contact information is:

| If you have any questions, suggestions of | r concerns <u>about your ri</u> g | ghts as a volunteer in this |
|---|---|---|
| research, contact the Institutional Review | Board at | or the Research Subject |
| Advocate at Wake Forest at | • | - |

#### Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you are an adolescent or young adult with cancer. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask


Adult Consent Form



the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to get feedback from providers on a new intervention to assess and address the needs of AYAs with cancer.

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY? 8 people will take part in this study.

#### WHAT IS INVOLVED IN THE STUDY?

You will participate in a 60-minute telephone interview. During this interview, we will ask you questions about your thoughts on NA-SB and how it might be implemented at you institution.

As part of this research study, you will be audiotaped. This is being for the purposes of transcription. You understand that you may request the recording be stopped at any time during the course of the research study. You can also withdraw your consent to use and disclose the audiotape before it is used. You should also understand that you will not be able to inspect, review, or approve the audiotapes before they are used in this study.

Please choose one of the following regarding the use and disclosure of the audiotape used in this research study:

\_\_\_\_\_ I would like the audiotapes of me to be destroyed once their use in this study is finished.

\_\_\_\_ The audiotapes of me can be kept for use in future studies provided they are kept secure and any future study will be reviewed by an IRB. I understand that I will not be able to inspect, review or approve their future use.

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for about <u>one day</u> (i.e., the time it takes to participate in 60-minute interview).

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

# WHAT ARE THE RISKS OF THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations

 Adult Consent Form



or tests. You should discuss the risk of being in this study with the study staff.

There is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

There are no expected direct benefits from taking part in the study.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to use NA-SB at your institution.

#### WHAT ARE THE COSTS?

All study costs, related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

#### WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Interview recordings from this study will be stored securely and only shared among members of the study team. They will be stored for approximately 6 months to allow for transcription and then permanently deleted. Note that, during interviews, participants can choose to stop the recording at any time.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

#### WILL YOU BE PAID FOR PARTICIPATING?

You will not be paid for participating.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by Wake Forest School of Medicine. The sponsor is providing money or other support to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you about your health or behaviors


Adult Consent Form



is considered <u>Protected Health Information</u>. The information we will collect for this research study includes **information about your physical**, **psychosocial**, **and practical needs**.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for at least six years after the study is finished. At that time any research information not already in your medical record will either be destroyed or it will be deidentified. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Sarah Birken that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:


Adult Consent Form



#### Sarah Birken



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

#### WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

You may choose not to take part or you may leave the study at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest or because the entire study has been stopped. Information about you may be removed from the study data and could be used for future research or shared with other researchers without additional consent from you.

By continuing, I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. I have had a chance to ask questions about being in this study and have those questions answered. By taking part in the study, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, <u>Sarah Birken, PhD</u> at or after-hours at .

Page **5** of **6**Adult Consent Form



The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at Research Subject Advocate at

You will be given a copy of this consent form.

 Adult Consent Form